CLINICAL TRIAL: NCT04338750
Title: Telephone Acceptance and Commitment Therapy Intervention for Caregivers of Adults With Alzheimer's Disease and Related Dementias (TACTICs): A Pilot Randomized Controlled Trial
Brief Title: Telephone Acceptance and Commitment Therapy Intervention for Caregivers of Adults With Dementia
Acronym: TACTICs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Indiana Clinical and Translational Sciences Institute (Other); Regenstrief Institute, Inc. (Other)
Responsible Party: Principal Investigator, Shelley Johns, Assistant Professor of Medicine, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2002468698
Record Dates: First submitted 2020-04-02; First posted 2020-04-08 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Anxiety; Anxiety Generalized; Anxiety Disorders and Symptoms; Caregiver Burnout
Keywords: Alzheimer's disease; Dementia; Caregiving; Caregiver; Anxiety; Acceptance and commitment therapy; Telehealth
MeSH Terms: conditions — Anxiety Disorders; Generalized Anxiety Disorder; Caregiver Burden; Alzheimer Disease; Dementia | interventions — Caregivers

STUDY DESIGN:
Intervention Model Description: Caregivers of adults with Alzheimer's disease or related dementias (N = 60) will be randomly assigned in equal numbers to Acceptance and Commitment Therapy delivered by telephone (TACTICs) or minimally-enhanced usual care (mEUC) using a block randomization scheme.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Principal Investigator and Outcomes Assessors are blinded to randomization sequence and randomization assignments for the duration of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telephone Acceptance and Commitment Therapy Intervention for Caregivers (TACTICs) (Experimental): Participants in the ACT arm will learn new and more adaptive ways to respond to challenges, including anxiety and the irreversibility of dementia and its behavioral manifestations.
  Interventions: Behavioral: Telephone Acceptance and Commitment Therapy Intervention for Caregivers
- minimally-Enhanced Usual Care (mEUC) (Active Comparator): Participants randomized to mEUC will receive educational, science-based reading and resources, including a listing of Alzheimer's Association sponsored support groups closest to their home address.
  Interventions: Behavioral: minimally-Enhanced Usual Care

INTERVENTIONS:
Behavioral: Telephone Acceptance and Commitment Therapy Intervention for Caregivers — Participants randomized to TACTICs will receive a manualized acceptance and commitment therapy intervention delivered via phone in 6 weekly 1-hour sessions by a trained Bachelor's-level interventionist. Participants in this intervention will practice various mindfulness exercises, clarify their values, and set specific goals consistent with their values. Sessions will incorporate discussion of patients' caregiving experiences. Through in-session and home practice of skills, participants will learn new and more adaptive ways to respond to anxiety and caregiving challenges. Participants will receive handouts on session topics and a CD with guided mindfulness practices.
  Other Names: TACTICs
  Arms: Telephone Acceptance and Commitment Therapy Intervention for Caregivers (TACTICs)
Behavioral: minimally-Enhanced Usual Care — Participants randomized to mEUC will receive a letter thanking them for participating in the trial along with the Alzheimer's Caregiving guide from the National Institute of Aging of the National Institutes of Health (https://www.nia.nih.gov/health/alzheimers/caregiving), coupled with a listing of the five Alzheimer's Association sponsored support groups closest to their home address.
  Other Names: mEUC
  Arms: minimally-Enhanced Usual Care (mEUC)

SUMMARY:
Caregivers of adults with dementia report higher distress, including anxiety and depressive symptoms, burden, and existential suffering, than caregivers of people with other chronic diseases. Acceptance and Commitment Therapy (ACT) is a behavioral intervention designed to increase psychological flexibility in the face of challenges. Results from our recent proof-of-concept study suggest that ACT is effective in reducing anxiety and associated psychological distress in dementia caregivers. In this study, we will randomize N=60 dementia caregivers in equal numbers to receive either 6 weekly 1-hour telephone-based ACT sessions (TACTICs; experimental) or minimally-enhanced usual care (mEUC; control). We hypothesize that our TACTICs intervention will be feasible and acceptable in this population and will have a greater impact on reducing anxiety and secondary outcomes from baseline to post-intervention, and 3 and 6 months later.

DETAILED DESCRIPTION:
The objective of this pilot randomized controlled trial is to assess feasibility, acceptability, and preliminary effects of Telephone Acceptance and Commitment Therapy Intervention for Caregivers (TACTICs) of adults with Alzheimer's disease or related dementias. Using a 2-arm randomized design, we will examine the effects of TACTICs compared to a minimally enhanced usual care group (mEUC) in N=60 dementia caregivers. Primary dementia caregivers with clinically-significant anxiety will be randomized in equal numbers to receive either TACTICs or mEUC. The specific aims are to: (1) Evaluate the feasibility and acceptability of TACTICs. Feasibility will be assessed using caregiver accrual, retention, and TACTICs session attendance rates. Acceptability will be assessed using a participant-reported satisfaction item administered upon intervention completion. (2) Measure the changes in caregiver anxiety and depressive symptoms, caregiver burden, wellbeing, and psychological flexibility at post-intervention (T2) and 3 months (T3) and 6 months (T4) post-intervention compared to baseline. Caregivers will be recruited from a variety of sources, including the Indiana Alzheimer's Disease Center (IADC), Aging Brain Care program at Eskenazi Health, and Indiana University Health geriatric psychiatry and neurology practices. Study staff will contact potentially-eligible caregivers to assess interest and verify eligibility. After providing informed consent and enrolling in the trial, interested and eligible caregivers will complete baseline measures and be randomly assigned in equal numbers to either the TACTICs intervention (n=30) or to mEUC (n=30) using a block randomization scheme. Randomization will be performed in REDCap using a SAS procedure. All study personnel will be blind to allocation sequence. The unblinded research coordinator will be responsible for randomizing participants in REDCap. The PI, Co-Investigators, and research assistants (i.e., recruiters and outcome assessors) will be blind to intervention assignment to reduce the risk of outcome expectancy bias and to enhance the rigor of the trial.

ELIGIBILITY:
Inclusion Criteria:

* 21 years or older
* Able to communicate in English
* Able to provide informed consent
* Listed as primary caregiver in the chart of a patient with Alzheimer's disease or a related dementia (ADRD)
* Self-identifies as ADRD patient's primary caregiver
* Intends to continue caregiving for ADRD patient for ≥12 months
* Clinically-elevated anxiety (score of 10 or higher on GAD-7)

Exclusion Criteria:

* Non-family member of the ADRD patient
* Has ADRD or other serious mental illness diagnosis such as bipolar or schizophrenia as determined by ICD-10 code

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-03-24 (Actual); Primary Completion 2021-04-09 (Actual); Study Completion 2021-04-09 (Actual)

PRIMARY OUTCOMES:
Change in Baseline Anxiety via Generalized Anxiety Disorder scale-7 (GAD-7) | baseline, post-intervention (7-9 weeks post-baseline), 3 months post-intervention, 6 months post-intervention
  Changes in anxiety will be measured using the Generalized Anxiety Disorder Scale (GAD-7), which contains 7 items with total scores ranging from 0 to 21. Scores of 5, 10, and 15 are cut-offs for mild, moderate, and severe anxiety, respectively. An add-on item assessing the patient's global impression of symptom-related impairment helps researchers understand the extent to which anxiety interferes in daily life. The GAD-7 has factorial validity for the diagnosis of general anxiety disorder and is sensitive to change.

SECONDARY OUTCOMES:
Change in Baseline Depressive Symptoms via Patient Health Questionnaire-9 (PHQ-9) | baseline, post-intervention (7-9 weeks post-baseline), 3 months post-intervention, 6 months post-intervention
  Changes in depressive symptoms will be measured using the 9-item Patient Health Questionnaire-9 (PHQ-9) to assess depressive symptoms. With total scores ranging from 0 to 27, scores of 5, 10, 15, and 20 represent mild, moderate, moderately severe, and severe depression, respectively. The PHQ-9 has factorial validity for the diagnosis of major depressive disorder.
Change in Baseline Caregiver Burden via Zarit Burden Interview (ZBI) | baseline, post-intervention (7-9 weeks post-baseline), 3 months post-intervention, 6 months post-intervention
  Changes in caregiver burden will be measured using the Zarit Burden Interview (ZBI). This two-factor, 22-item scale measures personal strain and role strain in caregiving by summing responses to a total score (0-20 little or no burden; 21-40 mild to moderate burden; 41-60 moderate to severe burden; and 61-88 severe burden). The ZBI measures change over time resulting from the progression of the patient's symptoms or from interventions aimed at reducing burden.
Change in Baseline Wellbeing via Experience of Suffering Scale (ESS) | baseline, post-intervention (7-9 weeks post-baseline), 3 months post-intervention, 6 months post-intervention
  Changes in wellbeing will be measured using the Experience of Suffering Scale (ESS). With prior testing in ADRD caregivers, the ESS contains 33 items across 3 subscales: physical (9 items), psychological (15 items), and existential (9 items) suffering. Total scores for each subscale are calculated with higher scores indicating more suffering within each domain.
Change in Baseline Coping via Brief COPE | baseline, post-intervention (7-9 weeks post-baseline), 3 months post-intervention, 6 months post-intervention
  Changes in coping will be measured with the 28-item Brief COPE, a measure of coping strategies used in response to stressors. Comprised of 28 coping strategies, the Brief COPE contains 14 two-item subscales, each analyzed separately: self-distraction, active coping, denial, substance use, use of emotional support, use of instrumental support, venting, behavioral disengagement, positive reframing, planning, humor, acceptance, religion, and self-blame.
Change in Baseline Psychological Flexibility via Acceptance and Action Questionnaire-II (AAQ-II) | baseline, post-intervention (7-9 weeks post-baseline), 3 months post-intervention, 6 months post-intervention
  Changes in psychological flexibility and its opposite, experiential avoidance, will be measured using the 7-item Acceptance and Action Questionnaire-II (AAQ-II). Respondents rate how true each statement (e.g., "It is okay if I remember something unpleasant") is for them on a 7-point Likert-type scale anchored from 1=never true to 7=always true. Higher scores indicate greater psychological flexibility or acceptance.
Change in Baseline Quality of Life via PROMIS Global Health measure | baseline, post-intervention (7-9 weeks post-baseline), 3 months post-intervention, 6 months post-intervention
  Changes in quality of life will be assessed with the 10-item PROMIS Global Health measure. On a 5-point scale, participants rate their mental and physical well-being with higher scores indicative of better health.
Change in Baseline Anticipatory Grief via Anticipatory Grief Scale (AGS) | baseline, post-intervention (7-9 weeks post-baseline), 3 months post-intervention, 6 months post-intervention
  Changes in anticipatory grief will be measured with the Anticipatory Grief Scale (AGS), a 27-item self-report tool designed to assess the bereavement experience of dementia caregivers. Items are scored on a 5-point Likert scale with responses ranging from "strongly disagree" to "strongly agree."

OTHER OUTCOMES:
Intervention feasibility: accrual rate | baseline
  We will assess the number of eligibly-screened caregivers who choose to consent and enroll in the trial. This accrual outcome speaks to intervention feasibility.
Intervention feasibility: attendance rate | post-intervention
  We will assess the total number of sessions that participants allocated to TACTICs attend (i.e., out of 6 sessions possible). This attendance outcome speaks to intervention feasibility.
Intervention feasibility: retention rate | 6 months post-intervention
  We will assess the number of enrolled subjects completing the final outcome assessment at 6 months post-intervention. This retention outcome speaks to intervention feasibility.
Intervention acceptability | post-intervention
  We will assess intervention acceptability using a brief investigator-created battery of quantitative and qualitative satisfaction items.
Health care and resource utilization | baseline, post-intervention, 3 months post-intervention, 6 months post-intervention
  Health care and resource utilization will be measured using an investigator-created battery of items. Items will assess caregiver-reported health and mental care utilization (e.g., ED, inpatient, outpatient) and services accessed or used to support their caregiving (e.g., support groups, respite care, in-home aid).

CONTACTS AND LOCATIONS:
Overall Officials: Shelley A. Johns, PsyD, Principal Investigator — Indiana University School of Medicine
Locations (1):
- Regenstrief Institute, Inc., Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: Yes
In future manuscripts, the authors will list contact information and state that IPD is available upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The data set will be made available to qualified investigators within 6 months of the publication of the primary outcome paper. Data will be available for at least 6 years.
Access Criteria: The data set and supporting information will be made available to qualified investigators to allow replication of analyses or secondary data analyses. The PI will review requests for data access. The investigators will be required to sign a data use agreement and obtain IRB approval before receiving the data set. The mechanism for data sharing will be reviewed by the IRB.